CLINICAL TRIAL: NCT07407764
Title: Exploratory Study of the Representations of the Inside of the Body of Adolescents With and Without Borderline Personality Disorder, Assessed Through a Drawing of the Inside of the Body, Interviews and Questionnaires.
Brief Title: Representations of the Body's Interior in Adolescence
Acronym: RICA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics committee refusal
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RICA
Record Dates: First submitted 2025-08-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adolescent - Emotional Problem; Personality Disorders in Adolescence; Body Representation; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Prospective, exploratory, descriptive and comparative study with cohorts. Qualitative study with a quantitative component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical cohort (Other): Adolescents with borderline personality disorder
  Interventions: Behavioral: Drawing of the inside of the body, interviews and questionnaires.
- Non-clinical cohort (Other): Adolescent without borderline personality disorder
  Interventions: Behavioral: Drawing of the inside of the body, interviews and questionnaires.

INTERVENTIONS:
Behavioral: Drawing of the inside of the body, interviews and questionnaires. — Use of various validated and non-validated tools to identify certain common characteristics, as well as more specific weaknesses, in the representations of the inside of the body of adolescents with no pathology, and adolescents with borderline personality disorder.

SUMMARY:
Representations of the inner body in adolescence: developmental characteristics and specificities in borderline personality disorders.

DETAILED DESCRIPTION:
The aim of this exploratory study is to describe the representations of the inside of the body of adolescents with borderline personality disorder, and adolescent without borderline personality disorder.

During an interview with a psychomotor specialist, participants will undergo tests, questionnaires and Internal body drawing test

ELIGIBILITY:
Inclusion Criteria:

* Non-clinical cohort :

  1. Adolescents aged 15 to 19
  2. High school students (seconde to terminale)
  3. Having signed a consent form to participate in the research, as well as their legal representative
  4. Affiliated to a social security regime
* Clinical cohort :

  1. Adolescents aged 15 to 19
  2. With a high school level (3rd year completed, transition to second year pronounced), whether enrolled or not.
  3. Having signed a consent form to participate in the research and their legal representative.
  4. Currently under psychiatric or pediatric care for psychiatric reasons.
  5. Diagnosed or suspected of having a borderline personality disorder,
  6. Affiliated to a social security regime

Exclusion Criteria:

Non-clinical cohort

1. Serious somatic pathology under treatment (e.g. cancer; recent or planned operations...)
2. Recognized sensory or neurological disability.
3. Known, diagnosed psychiatric pathologies (TCA, schizophrenia, etc.).
4. Refusal to participate by adolescent or parental guardians.

Clinical cohort :

1. Serious somatic pathology under treatment (e.g. cancer, recent or planned operations, etc.)
2. Recognized sensory or neurological disability.
3. Refusal to participate by adolescent or parental guardians.
4. Psychomotor assessment or follow-up by the researcher.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Type of organs represented | From enrollment to 2 months after enrollment
  Type of organs represented on drawing of body' s interior
Type of systems represented | From enrollment to 2 months after enrollment
  Type of systems represented on drawing of body' s interior
Number of organs represented | From enrollment to 2 months after enrollment
  Completeness of drawing of the inside of the body
Number of systems represented | From enrollment to 2 months after enrollment
  Completeness of drawing of the inside of the body + captions
Level of drawing elaboration | From enrollment to 2 months after enrollment
  Qualitative analyse of the drawing evaluated (complete and functional systems) - Minimum value: 0 (no elaboration / very simple drawing, incomplete or non-functional systems) Maximum value: 3 (high elaboration / detailed drawing with complete and functional systems) Interpretation: higher scores indicate a better outcome (higher level of drawing elaboration).

SECONDARY OUTCOMES:
Symbolic elements added to drawing | From enrollment to 2 months after enrollment
  Describe "non-anatomical" themes added to the drawing
Type of anatomical errors in the drawing | From enrollment to 2 months after enrollment
  Describe anatomical errors in the drawing
Scores obtained from questionnaires: Multidimensional Assessment of Interoceptive Awareness):Interoceptive awareness, | From enrollment to 2 months after enrollment
  Demonstrate alterations in various dimensions in borderline adolescents
Scores obtained from questionnaires: Postural Awareness Scale_Proprioceptive awareness, | From enrollment to 2 months after enrollment
  Demonstrate alterations in various dimensions in borderline adolescents
Scores obtained from questionnaires: Toronto Alexithymia Scale-20)_Emotional awareness (degree of alexithymia) | From enrollment to 2 months after enrollment
  Demonstrate alterations in various dimensions in borderline adolescents
Scores obtained from questionnaires: Body Image Questionnaire_Body satisfaction | From enrollment to 2 months after enrollment
  Demonstrate alterations in various dimensions in borderline adolescents
Frequency of responses to questions about drawing the inside of the body | From enrollment to 2 months after enrollment
  Gather participants' opinions on the proposed inner-body drawing test
Type of symbolic representations emerging through the interview | From enrollment to 2 months after enrollment
  Evaluate symbolic representations of the body through language.
Frequency of responses to additional questions about the body's interior | From enrollment to 2 months after enrollment
  Evaluate participants' level of preoccupation with and experience of the inner body.
Questionnaire scores by age | From enrollment to 2 months after enrollment
  To explore differences attributable to the developmental aspect of representations of the body's interior: 30 control high school students (RICA)/200 young adult students and adult students over 25 (results obtained in a preliminary study).